CLINICAL TRIAL: NCT04763954
Title: The Effect of a Therapeutic Game With or Without Email Coaching in Improving the Emotional Abilities in Students
Brief Title: Guided and Unguided Therapeutic Game to Improve Emotional Abilities of Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Cristina Lorint, Ph.D Student, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1396/ 10.02.2021
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Emotional Stress
Keywords: emotional skills; emotional abilities; stress; relaxation
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Game and control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Game (Experimental): Group that receives the game intervention (the trial version and the access to level 2 and level 7
  Interventions: Other: Rethink therapeutic game
- Control (No Intervention): Group without intervention
- Guidance (Experimental): Group that receives the game (the same levels as group 1) and email coaching one day after completing the game.
  Interventions: Other: Rethink therapeutic game

INTERVENTIONS:
Other: Rethink therapeutic game — The Rethink therapeutic game is a 7 levels online game developed and tested for children. Each level is based on a specific skill and its efficiency has been previously studies in children.
  Arms: Game; Guidance

SUMMARY:
The aim of the study is to investigate the efficiency of a therapeutic online game, with and without coaching, in training emotional abilities of students.

DETAILED DESCRIPTION:
The study is a randomized control trial with three groups. We will perform measurements before the intervention, after the intervention and at one month follow-up.

Participants will be students and will be randomized into three groups using a randomization program. The first group will be the gaming with coaching group, the second group will bw the gaming without coaching group and the third group will be the control group.

Measurements will be performed before receiving the game, after the intervention and at one month follow-up. We will measure depression, anxiety, stress and well-being as primary outcomes, solution focus orientation as secondary outcome and rational and irrational cognitions as mechanism outcome. All questionnaires will be completed online in a Google Form.

The intervention will consist of the Rethink game. Rethink is a therapeutic game developed and tested to improve emotional abilities in children. Participants in our study will test two levels of Rethink as well as a trial version of the game. Each level of the game is focused on a component:

* Level 1: recognition of emotions
* Level 2: relaxation and mindfulness
* Level 3: rational and irrational cognitions
* Level 4:changing the cognitions
* Level 5: problem-solving
* Level 6: positive emotions
* Level 7: summary of previous aqusitions

ELIGIBILITY:
Inclusion Criteria:

* being a student in a public or private university from Romania

Exclusion Criteria:

* not being enrolled as a student in a university from Romania

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Baseline emotions | Pre-intervention (one day before the intervention)
  Measured with Profile of Emotional Distress
Emotions after intervention in a stressful condition | Post-intervention - before a stressful event (before an exam)
  Measured with Profile of Emotional Distress
Changes in time in emotions after intervention | Post-intervention at one month after the intervention
  Measured with Profile of Emotional Distress

SECONDARY OUTCOMES:
Baseline cognitions | Pre-intervention (one day before the intervention)
  Measured with Attitudinal Beliefs Scale
Cognitions after intervention in stress condition | Post-intervention - before a stressful event (before an exam)
  Measured with Attitudinal Beliefs Scale
Changes in time in cognitions after intervention | Post-intervention at one month after the intervention
  Measured with Attitudinal Beliefs Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cristinalorint@Psychology.Ro, Cluj-Napoca, Cluj, Romania

REFERENCES:
- [Derived] Tomoiaga C, David O. The Efficacy of Guided and Unguided Game-Based Cognitive-Behavioral Therapy in Reducing Distress in College Students. Games Health J. 2022 Sep 6. doi: 10.1089/g4h.2021.0195. Online ahead of print. PMID 36067336